CLINICAL TRIAL: NCT00996216
Title: An Open-label, Multi-centre Rollover Study to Assess the Safety and Efficacy of Eltrombopag in Thrombocytopenic Subjects With Hepatitis C Virus (HCV) Infection Who Are Otherwise Eligible to Initiate Antiviral Therapy (Peginterferon Alfa-2a or Peginterferon Alfa-2b Plus Ribavirin)
Brief Title: Clinical Trial for Non-responders Who Previously Participated in Eltrombopag Studies TPL 103922 or TPL 108390
Acronym: ENABLE-ALL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 108392
Record Dates: First submitted 2009-10-01; First posted 2009-10-16 (Estimated); Results first posted 2013-12-06 (Estimated); Last update posted 2013-12-06 (Estimated); Status verified 2013-08

CONDITIONS: Hepatitis C
Keywords: Peginterferon; Platelets; Ribavirin; Hepatitis C-related thrombocytopenia; Thrombocytopenia; Hepatitis C; Thrombopoietin
MeSH Terms: conditions — Hepatitis C; Thrombocytopenia; Jacobs syndrome | interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open-label eltrombopag (Experimental): Open-label eltrombopag with dose titrations to support adequate platelet counts.
  Interventions: Drug: Eltrombopag; Drug: Antiviral therapy

INTERVENTIONS:
Drug: Eltrombopag — Eltrombopag starting at 25 mg dose and titrated in Part 1 of study to 50, 75, 100 mg. Platelet count must reach sufficient level to allow initiation of antiviral therapy. Eltrombopag dose may be adjusted during antiviral treatment phase of study to maintain platelet count to continue antiviral therapy without adjustment to antiviral dose.
  Other Names: Promacta
Drug: Antiviral therapy — Combination of either peginterferon alfa-2a or alfa-2b with ribavirin at investigator's discretion.

SUMMARY:
The purpose of this study is to test the safety and tolerability of eltrombopag when used to increase and maintain platelet count. Platelet count to be maintained at a level sufficient to facilitate initiation of antiviral therapy, to minimize antiviral therapy dose reductions, and to avoid permanent discontinuation of antiviral therapy.

ELIGIBILITY:
Inclusion Criteria:

* Prior participation in protocol TPL103922 or TPL108390 and completed the Week 24 Follow Up Visit in TPL103922 or TPL108390
* Male or female ≥18 years old
* Evidence of chronic HCV infection
* While participating in TPL103922 or TPL108390, discontinued from study drug due to thrombocytopenia
* Appropriate candidate for antiviral therapy with pegylated interferon plus ribavirin
* Platelet count <75,000
* Fertile males and females must use two forms of effective contraception during treatment and for 24 weeks after treatment
* Ability to understand and comply with the protocol requirements and instructions
* Ability to provide written informed consent

Exclusion Criteria:

* Decompensated liver disease
* Known hypersensitivity, intolerance, or allergy to interferon, ribavirin, eltrombopag, or their ingredients
* History of clinically significant bleeding from oesophageal or gastric varices
* History of arterial or venous thrombosis and two or more of the following risk factors: hereditary thrombophilic disorders; hormone replacement therapy; systemic contraception (containing estrogen); smoking; diabetes; hypercholesterolemia; medication for hypertension or cancer
* Pre-existing cardiac disease (congestive heart failure Grade III/IV) or arrhythmias known to involve the risk of thromboembolic events (e.g. atrial fibrillation)
* Evidence of hepatocellular carcinoma
* HIV or Hepatitis B infection
* Therapy with anti-neoplastic or immunomodulatory treatment within six months prior to eltrombopag therapy
* Malignancy diagnosed or treated within the past five years. Except for localized basal or squamous cell carcinoma treated by local excision or malignancies that were adequately treated and, in the opinion of the oncologist, have an excellent chance of cancer-free survival.
* Pregnant or nursing women
* Men with a female partner who is pregnant
* History of alcohol/drug abuse or dependence within six months of the study start unless participating in a controlled rehabilitation programme.
* Treatment with an investigational drug or interferon within 30 days or 5 half-lives (whichever is longer) of the screening visit
* History or platelet clumping that prevents reliable measurement of platelet counts
* Evidence of portal vein thrombosis within three months of baseline visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-09; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (28):
- United States (6):
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Honolulu, Hawaii
  - GSK Investigational Site, Manhasset, New York
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Seattle, Washington
- Australia (3):
  - GSK Investigational Site, Camperdown, New South Wales
  - GSK Investigational Site, Randwick, New South Wales
  - GSK Investigational Site, Herston, Queensland
- Canada (2):
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- France (3):
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Pessac
- Germany (5):
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Ulm, Baden-Wurttemberg
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Düsseldorf, North Rhine-Westphalia
  - GSK Investigational Site, Berlin, State of Berlin
- GSK Investigational Site, Athens, Greece
- Italy (3):
  - GSK Investigational Site, Bologna, Emilia-Romagna
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Milan, Lombardy
- GSK Investigational Site, Lahore, Pakistan
- Spain (4):
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Pontevedra
  - GSK Investigational Site, Valencia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10^9 cells (Giga) per liter=Gi/L; participants=par.; polyethylene glycol=Peg; interferon=INF.
Pre-assignment Details: In Part (P) 1, the treatment goal was to increase the platelet count to >=90 Gi/L. In P 2, par. continued on the selected P 1 dose of eltrombopag (dose effectively raising platelets to >=90 or >=100 Gi/L). Eltrombopag was given in combination with antiviral therapy (Peg INF alfa-2a or Peg INF alfa-2b and ribavirin) for the duration of treatment.
Groups:
- Eltrombopag: In the Pre-antiviral Treatment Phase, participants (par.) with a platelet count of <75000/microliter (µL) received eltrombopag once daily for a minimum of 2 weeks and a maximum of 9 weeks in sequential dose escalations (25 milligrams [mg] for a minimum of 2 weeks, 50 mg for 1-2 weeks, 75 mg for 1-2 weeks, and 100 mg for 1-3 weeks) until platelet counts reached either >=90000/µL or 100000/µL. Par. who achieved the desired platelet count continued with eltrombopag in Part 2 along with antiviral treatment. Par. who did not achieve the desired platelet count completed the follow-up visits and were withdrawn from the study. Once the desired platelet counts were reached in Part 1 (>=90 Gi/L or >=100 Gi/L), par. continued to receive the dose of eltrombopag from Part 1 and polyethylene glycol (Peg) interferon (INF) alfa-2a (>=90 Gi/L) or Peg IFN alfa-2b (>=100 Gi/L) plus ribavirin. Dose adjustments of eltrombopag were permitted to achieve and maintain an appropriate platelet count.
Period: Part 1 (Pre-Antiviral Treatment Phase)
Arm/Group | Eltrombopag
Started | 27
Completed | 26
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Part 2 (Antiviral Treatment Phase)
Arm/Group | Eltrombopag
Started | 25 (One participant who completed Part 1 didn't qualify to begin antiviral treatment in Part 2.)
Completed | 21
Not Completed | 4
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Eltrombopag
Number analyzed (Participants) | 27
Age Continuous [Mean (Standard Deviation); unit: Years] | 51.3 (7.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 20
Race/Ethnicity, Customized [Number; unit: participants]
  Central/South Asian Heritage | 2
  White | 25

OUTCOME MEASURES:

1. Secondary Outcome: Platelet Counts at the Indicated Time Points
Description: Blood samples were collected for the measurement of platelet count. For each participant, the duration of Part 1 treatment varies between 2 and 9 weeks.
Time Frame: From the start of investigational product up to the 24-week follow-up visit after the last dose in Part 2 or early withdrawal (up to 96 weeks)
Population: Pre-antiviral Safety Population
Measure: Mean (Standard Deviation); unit: Gi/L
Arm/Group | Eltrombopag
Number analyzed (Participants) | 27
Gi/L
  Screening, n=27 | 53.1 (12.90)
  Part 1/Day 1, n=27 | 55.9 (18.69)
  Part 1/Week 1, n=25 | 73.3 (29.27)
  Part 1/Week 2, n=16 | 83.2 (27.90)
  Part 1/Week 3, n=8 | 73.4 (26.53)
  Part 1/Week 4, n=7 | 75.6 (19.95)
  Part 1/Week 5, n=5 | 72.2 (18.29)
  Part 1/Week 6, n=5 | 81.6 (14.45)
  Part 1/Week 7, n=5 | 76.2 (19.88)
  Part 1/Week 8, n=3 | 91.7 (22.81)
  Part 2/Antiviral Baseline, n=25 | 132.9 (33.72)
  Part 2/Week 1, n=25 | 106.7 (37.80)
  Part 2/Week 2, n=25 | 93.2 (42.98)
  Part 2/Week 4, n=23 | 80.5 (30.64)
  Part 2/Week 8, n=21 | 80.3 (24.40)
  Part 2/Week 12, n=20 | 83.1 (31.72)
  Part 2/Week 16, n=16 | 85.8 (27.61)
  Part 2/Week 20, n=14 | 75.3 (22.54)
  Part 2/Week 24, n=11 | 78.6 (30.63)
  Part 2/Week 28, n=9 | 90.3 (50.09)
  Part 2/Week 32, n=7 | 86.1 (72.12)
  Part 2/Week 36, n=6 | 76.8 (53.77)
  Part 2/Week 40, n=5 | 55.8 (27.65)
  Part 2/Week 44, n=5 | 54.4 (29.18)
  Part 2/Week 48, n=2 | 68.0 (29.70)
  Part 2/Week 52, n=1 | 49.0 (NA) — A standard deviation cannot be calculated when mean data are available for only one participant.
  Part 2/Week 56, n=1 | 47.0 (NA) — A standard deviation cannot be calculated when mean data are available for only one participant.
  Part 2/Week 60, n=1 | 43.0 (NA) — A standard deviation cannot be calculated when mean data are available for only one participant.
  Part 2/Week 64, n=1 | 43.0 (NA) — A standard deviation cannot be calculated when mean data are available for only one participant.
  Part 2/Week 68, n=1 | 44.0 (NA) — A standard deviation cannot be calculated when mean data are available for only one participant.
  Post-treatment/4 Week Follow-up, n=23 | 77.8 (33.48)
  Post-treatment/24 Week Follow-up, n=22 | 52.5 (17.91)
  Investigational product discontinuation, n=26 | 91.3 (38.78)
  Maximum value post-Baseline, n=26 | 145.5 (43.68)

2. Secondary Outcome: Number of Particpants Who Initiated Antiviral Therapy
Description: The number of participants who completed the Pre-antiviral Phase (Part 1) and proceeded to the Antiviral Phase (Part 2) are summarized.
Time Frame: From the start of the investigational product up to 9 weeks (median of 21 days)
Population: Pre-antiviral Safety Population
Measure: Number; unit: Participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 27
Participants
  Yes | 25
  No | 2

3. Primary Outcome: Number of Participants With Any Adverse Event (AE) and Any Serious Adverse Event (SAE) in Part 1
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, may jeopardize the participant or require medical or surgical intervention to prevent one of the other outcomes listed, or is an event of possible drug-induced liver injury. Refer to the general AE/SAE module for a list of AEs and SAEs.
Time Frame: From the start of investigational product up to the start of antiviral therapy (up to 9 weeks; median of 21 days)
Population: Pre-antiviral Safety Population: all participants who received study drug in the Pre-antiviral Treatment Phase (Part 1) of the study
Measure: Number; unit: Participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 27
Participants
  Any SAE | 0
  Any AE | 9

4. Primary Outcome: Number of Participants With Any AE and Any SAE in Part 2
Description: as for outcome 3
Time Frame: From the date of initiation of antiviral therapy (Antiviral Baseline Visit [between Study Day 14 and Study Day 65]) to the completion of the follow-up period (up to Week 96/WD)
Population: Antiviral Safety Population: all participants who entered the Antiviral Treatment Phase (Part 2) of the study and who received at least one dose of antiviral therapy
Measure: Number; unit: Participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 25
Participants
  Any SAE | 5
  Any AE | 25

5. Primary Outcome: Number of Participants With the Indicated Worst-case Division of Acquired Immune Deficiency Syndrome (DAIDS) Grade Increases From Screening for the Indicated Clinical Chemistry Parameters During Part 1
Description: Blood samples were collected for the measurement of clinical chemistry parameters. The DAIDS grades are utilized for measuring the severity of AEs. Grade 1, mild; Grade 2, moderate; Grade 3, severe; Grade 4, potentially life threatening.
Time Frame: From Screening up to the start of antiviral therapy (up to 9 weeks; median of 21 days)
Population: Pre-antiviral Safety Population. Only participants with data available at the specified time point were analyzed.
Measure: Number; unit: Participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 26
Participants
  Alanine amino transferase, Any Increase | 2
  Alanine amino transferase, Increase to Grade 1 | 1
  Alanine amino transferase, Increase to Grade 2 | 0
  Alanine amino transferase, Increase to Grade 3 | 1
  Alanine amino transferase, Increase to Grade 4 | 0
  Albumin, Any Increase | 1
  Albumin, Increase to Grade 1 | 1
  Albumin, Increase to Grade 2 | 0
  Albumin, Increase to Grade 3 | 0
  Albumin, Increase to Grade 4 | 0
  Alkaline phosphatase, Any Increase | 1
  Alkaline phosphatase, Increase to Grade 1 | 1
  Alkaline phosphatase, Increase to Grade 2 | 0
  Alkaline phosphatase, Increase to Grade 3 | 0
  Alkaline phosphatase, Increase to Grade 4 | 0
  Aspartate amino transferase, Any Increase | 2
  Aspartate amino transferase, Increase to Grade 1 | 2
  Aspartate amino transferase, Increase to Grade 2 | 0
  Aspartate amino transferase, Increase to Grade 3 | 0
  Aspartate amino transferase, Increase to Grade 4 | 0
  Creatinine, Any Increase | 0
  Creatinine, Increase to Grade 1 | 0
  Creatinine, Increase to Grade 2 | 0
  Creatinine, Increase to Grade 3 | 0
  Creatinine, Increase to Grade 4 | 0
  Total bilirubin, Any Increase | 10
  Total bilirubin, Increase to Grade 1 | 6
  Total bilirubin, Increase to Grade 2 | 4
  Total bilirubin, Increase to Grade 3 | 0
  Total bilirubin, Increase to Grade 4 | 0
  Uric acid, Any Increase | 3
  Uric acid, Increase to Grade 1 | 3
  Uric acid, Increase to Grade 2 | 0
  Uric acid, Increase to Grade 3 | 0
  Uric acid, Increase to Grade 4 | 0

6. Primary Outcome: Number of Participants With the Indicated Worst-case DAIDS Grade Increases From the Antiviral Baseline Visit for the Indicated Clinical Chemistry Parameter During Part 2
Description: as for outcome 5
Time Frame: From Day 0 of Part 2 (Antiviral Baseline Visit [between Study Day 14 and Study Day 65) to the completion of the follow-up period (up to Week 96/WD)
Population: Antiviral Safety Population
Measure: Number; unit: Participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 25
Participants
  Alanine amino transferase, Any Increase | 4
  Alanine amino transferase, Increase to Grade 1 | 3
  Alanine amino transferase, Increase to Grade 2 | 0
  Alanine amino transferase, Increase to Grade 3 | 1
  Alanine amino transferase, Increase to Grade 4 | 0
  Albumin, Any Increase | 9
  Albumin, Increase to Grade 1 | 4
  Albumin, Increase to Grade 2 | 5
  Albumin, Increase to Grade 3 | 0
  Albumin, Increase to Grade 4 | 0
  Alkaline phosphatase, Any Increase | 7
  Alkaline phosphatase, Increase to Grade 1 | 7
  Alkaline phosphatase, Increase to Grade 2 | 0
  Alkaline phosphatase, Increase to Grade 3 | 0
  Alkaline phosphatase, Increase to Grade 4 | 0
  Aspartate amino transferase, Any Increase | 9
  Aspartate amino transferase, Increase to Grade 1 | 1
  Aspartate amino transferase, Increase to Grade 2 | 8
  Aspartate amino transferase, Increase to Grade 3 | 0
  Aspartate amino transferase, Increase to Grade 4 | 0
  Creatinine, Any Increase | 1
  Creatinine, Increase to Grade 1 | 0
  Creatinine, Increase to Grade 2 | 0
  Creatinine, Increase to Grade 3 | 1
  Creatinine, Increase to Grade 4 | 0
  Total bilirubin, Any Increase | 16
  Total bilirubin, Increase to Grade 1 | 1
  Total bilirubin, Increase to Grade 2 | 5
  Total bilirubin, Increase to Grade 3 | 10
  Total bilirubin, Increase to Grade 4 | 0
  Uric acid, Any Increase | 5
  Uric acid, Increase to Grade 1 | 4
  Uric acid, Increase to Grade 2 | 1
  Uric acid, Increase to Grade 3 | 0
  Uric acid, Increase to Grade 4 | 0

7. Primary Outcome: Number of Participants With the Indicated Worst-case DAIDS Grade Increases From Screening for the Indicated Hematology Parameters During Part 1
Description: Blood samples were collected for the measurement of hematology parameters. The DAIDS grades are utilized for measuring the severity of AEs. Grade 1, mild; Grade 2, moderate; Grade 3, severe; Grade 4, potentially life threatening.
Time Frame: From Screening up to the start of antiviral therapy (up to 9 weeks; median of 21 days)
Population: Pre-antiviral Safety Population. Only participants with data available at the specified time point were analyzed.
Measure: Number; unit: Participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 26
Participants
  Hemoglobin, Any Increase | 2
  Hemoglobin, Increase to Grade 1 | 2
  Hemoglobin, Increase to Grade 2 | 0
  Hemoglobin, Increase to Grade 3 | 0
  Hemoglobin, Increase to Grade 4 | 0
  Lymphocytes, Any Increase | 3
  Lymphocytes, Increase to Grade 1 | 1
  Lymphocytes, Increase to Grade 2 | 1
  Lymphocytes, Increase to Grade 3 | 1
  Lymphocytes, Increase to Grade 4 | 0
  Total neutrophils, Any Increase | 3
  Total neutrophils, Increase to Grade 1 | 3
  Total neutrophils, Increase to Grade 2 | 0
  Total neutrophils, Increase to Grade 3 | 0
  Total neutrophils, Increase to Grade 4 | 0
  White Blood cell count, Any Increase | 2
  White Blood cell count, Increase to Grade 1 | 0
  White Blood cell count, Increase to Grade 2 | 2
  White Blood cell count, Increase to Grade 3 | 0
  White Blood cell count, Increase to Grade 4 | 0

8. Primary Outcome: Number of Participants With the Indicated Worst-case DAIDS Grade Increases From the Antiviral Baseline Visit for the Indicated Hematology Parameters During Part 2
Description: Blood samples were collected for the measurement of hematology chemistry parameters. The DAIDS grades are utilized for measuring the severity of AEs. Grade 1, mild; Grade 2, moderate; Grade 3, severe; Grade 4, potentially life threatening.
Time Frame: as for outcome 6
Population: Antiviral Safety Population
Measure: Number; unit: Participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 25
Participants
  Hemoglobin, Any Increase | 12
  Hemoglobin, Increase to Grade 1 | 1
  Hemoglobin, Increase to Grade 2 | 5
  Hemoglobin, Increase to Grade 3 | 5
  Hemoglobin, Increase to Grade 4 | 1
  Lymphocytes, Any Increase | 15
  Lymphocytes, Increase to Grade 1 | 1
  Lymphocytes, Increase to Grade 2 | 3
  Lymphocytes, Increase to Grade 3 | 3
  Lymphocytes, Increase to Grade 4 | 8
  Total neutrophils, Any Increase | 23
  Total neutrophils, Increase to Grade 1 | 4
  Total neutrophils, Increase to Grade 2 | 10
  Total neutrophils, Increase to Grade 3 | 8
  Total neutrophils, Increase to Grade 4 | 1
  White Blood Cell count, Any Increase | 20
  White Blood Cell count, Increase to Grade 1 | 5
  White Blood Cell count, Increase to Grade 2 | 7
  White Blood Cell count, Increase to Grade 3 | 7
  White Blood Cell count, Increase to Grade 4 | 1

9. Primary Outcome: Number of Participants With a Decrease in Visual Acuity During Parts 1 and 2
Description: Visual acuity (VA) is defined as acuteness or clearness of vision.
Time Frame: as for outcome 1
Population: Entire Safety Population: all participants in the Pre-antiviral Safety Population
Measure: Number; unit: Participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 27
Participants
  Decrease in Visual Acuity, Yes | 10
  Decrease in Visual Acuity, No | 15
  Decrease in Visual Acuity, Missing or Unknown | 2

10. Primary Outcome: Number of Participants With the Indicated Change in logMAR Scale Values During Parts 1 and 2
Description: LogMAR (logarithm of the minimum angle of resolution) charts are used to measure an individual's visual acuity. LogMAR, expressed as the (decadic) logarithm of the minimum angle of resolution (range from +1.00 to -0.30), converts the geometric sequence of a traditional chart to a linear scale. As there are 5 letters per line, the total score for a line on the LogMAR chart represents a change of 0.1 log units.
Time Frame: as for outcome 1
Population: Entire Safety Population
Measure: Number; unit: Participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 27
Participants
  logMAR Changes, <0.10 (No Change or Improvement) | 15
  logMAR Changes, >=0.10 to <0.20 (Loss of 1 Line) | 6
  logMAR Changes, >=0.20 to <0.30 (Loss of 2 Lines) | 3
  logMAR Changes, >=0.30 (Loss of 3 Lines or more) | 1
  logMAR Changes, Missing or Unknown | 2

11. Primary Outcome: Number of Participants With a logMAR Change >=0.15 During Parts 1 and 2
Description: as for outcome 10
Time Frame: as for outcome 1
Population: Entire Safety Population
Measure: Number; unit: Participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 27
Participants
  logMAR change, Yes | 4
  logMAR change, No | 21
  logMAR change, Missing or Unknown | 2

12. Secondary Outcome: Number of Participants Achieving Antiviral Treatment Milestones of Sustained Virological Response (SVR), Rapid Virological Response (RVR), Early Virological Response (EVR), and End of Treatment Response (ETR)
Description: SVR is defined as non-detectable Hepatitis C virus (HCV) ribonucleic acid (RNA) at 24 weeks post-completion of the planned treatment period (i.e., Week 48 or 72 for genotype 2/3 or Week 72 for non-genotype 2/3). RVR is defined as undetectable HCV RNA after 4 weeks of antiviral treatment. EVR is defined as clinically significant reduction in HCV RNA (>=2 log10 drop or undetectable) after 12 weeks of antiviral treatment. ETR is defined as undetectable HCV RNA at the end of antiviral treatment.
Time Frame: From the start of investigational product in Part 2 up to the 24-week follow-up visit after the last dose in Part 2 or early withdrawal (up to 96 weeks)
Population: Antiviral Safety Population. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles). Different participants may have been analyzed for different parameters, so the overall number of participants analyzed reflects everyone in the Antiviral Safety Population.
Measure: Number; unit: Participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 25
Participants
  SVR, Yes, n=17 | 4
  SVR, No, n=17 | 13
  RVR, Yes, n=12 | 3
  RVR, No, n=12 | 9
  EVR, Yes, n=15 | 15
  EVR, No, n=15 | 0
  ETR, Yes, n=21 | 9
  ETR, No, n=21 | 12

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of study medication until the end of the 24-week follow up period (up to Week 96/WD).
Groups:
- Eltrombopag (Part 1): In the Pre-antiviral Treatment Phase, participants (par.) with a platelet count of <75000/microliter (µL) received eltrombopag once daily for a minimum of 2 weeks and a maximum of 9 weeks in sequential dose escalations (25 milligrams [mg] for a minimum of 2 weeks, 50 mg for 1-2 weeks, 75 mg for 1-2 weeks, and 100 mg for 1-3 weeks) until platelet counts reached either >=90000/µL or 100000/µL. Par. who achieved the desired platelet count continued with eltrombopag in Part 2 along with antiviral treatment. Par. who did not achieve the desired platelet count completed the follow-up visits and were withdrawn from the study.
- Eltrombopag (Part 2): Once the desired platelet counts were reached in Part 1 (>=90 Gi/L or >=100 Gi/L), par. continued to receive the dose of eltrombopag from Part 1 and polyethylene glycol (Peg) interferon (INF) alfa-2a (>=90 Gi/L) or Peg IFN alfa-2b (>=100 Gi/L) plus ribavirin. Dose adjustments of eltrombopag were permitted to achieve and maintain an appropriate platelet count.
Arm/Group | Eltrombopag (Part 1) | Eltrombopag (Part 2)
Serious Adverse Events (participants affected / at risk) | 0/27 | 5/25
Other Adverse Events (participants affected / at risk) | 9/27 | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag (Part 1) (N=27) | Eltrombopag (Part 2) (N=25)
Hepatic encephalopathy (Nervous system disorders) | 0 | 1
Myoclonic epilepsy (Nervous system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Metabolic disorder (Metabolism and nutrition disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag (Part 1) (N=27) | Eltrombopag (Part 2) (N=25)
Nausea (Gastrointestinal disorders) | 2 | 7
Abdominal distension (Gastrointestinal disorders) | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 3
Constipation (Gastrointestinal disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 2
Flatulence (Gastrointestinal disorders) | 1 | 1
Varices oesophageal (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 4
Vomiting (Gastrointestinal disorders) | 0 | 4
Ascites (Gastrointestinal disorders) | 0 | 3
Haematemesis (Gastrointestinal disorders) | 0 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Faeces discoloured (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Hypertrophy of tongue papillae (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 7
Parkinsonism (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 2
Disturbance in attention (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1
Hyperaesthesia (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1
Myoclonic epilepsy (Nervous system disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 6
Neutropenia (Blood and lymphatic system disorders) | 1 | 3
Leukopenia (Blood and lymphatic system disorders) | 0 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 4
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 2
Viral rhinitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 4
Upper respiratory tract infection (Infections and infestations) | 0 | 3
Candidiasis (Infections and infestations) | 0 | 2
Cellulitis (Infections and infestations) | 0 | 1
Ear infection (Infections and infestations) | 0 | 1
Furuncle (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1
Urinary tract infection bacterial (Infections and infestations) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 5
Pyrexia (General disorders) | 0 | 9
Fatigue (General disorders) | 0 | 7
Influenza like illness (General disorders) | 0 | 5
Chills (General disorders) | 0 | 3
Irritability (General disorders) | 0 | 2
Oedema (General disorders) | 0 | 2
Oedema peripheral (General disorders) | 0 | 2
Chest pain (General disorders) | 0 | 1
Injection site erythema (General disorders) | 0 | 1
Injection site pruritus (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 3
Sleep disorder (Psychiatric disorders) | 0 | 2
Aggression (Psychiatric disorders) | 0 | 1
Anger (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Depressed mood (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Mood swings (Psychiatric disorders) | 0 | 1
Nervousness (Nervous system disorders) | 0 | 1
Vision blurred (Eye disorders) | 0 | 2
Cataract (Eye disorders) | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 1
Eye discharge (Eye disorders) | 0 | 1
Retinal exudates (Eye disorders) | 0 | 1
Retinal haemorrhage (Eye disorders) | 0 | 1
Retinopathy (Eye disorders) | 0 | 1
Visual acuity reduced (Eye disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 2
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Nocturia (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Metabolic disorder (Metabolism and nutrition disorders) | 0 | 1
Haematoma (Vascular disorders) | 0 | 2
Pallor (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 0 | 1
Testicular pain (Reproductive system and breast disorders) | 0 | 2
Hepatic pain (Hepatobiliary disorders) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.